CLINICAL TRIAL: NCT00520442
Title: Ibuprofen Versus Acetaminophen With Codeine In Acute Pediatric Forearm Fractures
Brief Title: Acute Pediatric Fracture Analgesia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fracture Pain
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Fracture
Keywords: fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Ibuprofen; Acetaminophen; Codeine; Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental)
  Interventions: Drug: ibuprofen
- acetamin w codeine (Active Comparator)
  Interventions: Drug: acetamin w codeine

INTERVENTIONS:
Drug: ibuprofen
  Other Names: motrin; advil
  Arms: Ibuprofen
Drug: acetamin w codeine
  Other Names: tylenol with codeine, T3
  Arms: acetamin w codeine

SUMMARY:
A clinical trial comparing ibuprofen and acetaminophen with codeine for children after discharge from the emergency department. We hypothesize that Ibuprofen will provide 20% more effective analgesia compared to acetaminophen with codeine in children with uncomplicated forearm fractures.

DETAILED DESCRIPTION:
A clinical trial comparing ibuprofen and acetaminophen with codeine for children after discharge from the emergency department. We hypothesize that Ibuprofen will provide 20% more effective analgesia compared to acetaminophen with codeine in children with uncomplicated forearm fractures. A random table will be used to generate an assignment of the participants to either ibuprofen or acetaminophen with codeine. Assessment of the child's pain severity, pain medication use, functional limitations and parental satisfaction will allow for identification of a difference in the management of pain in the first 72 hours after a forearm fracture. Descriptive statistics will be used to analyze demographic data.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 4-18 years of age with an uncomplicated forearm fracture that is evaluated within 12 hours of injury and requires only splinting

Exclusion Criteria:

* A history of a bleeding disorder, uncontrolled chronic medical disease, regularly use of or allergy to acetaminophen, ibuprofen, or codeine or developmental delay

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 335 (Estimated)
Dates: Start 2003-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change to rescue medication | First 72 hours after ED discharge

SECONDARY OUTCOMES:
Pain score | First 72 hours after ED discharge
Functional outcomes: eat, sleep, play, school | First 72 hours after ED discharge

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drendel, DO, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States